CLINICAL TRIAL: NCT04926415
Title: Effects of Transcutaneous Auricular Vagus Nerve Stimulation on Obesity and Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burrell College of Osteopathic Medicine (Other)
Responsible Party: Principal Investigator, Harald Stauss, Associate Professor of Pharmacology, Burrell College of Osteopathic Medicine
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 0079_2021
Record Dates: First submitted 2021-06-02; First posted 2021-06-15 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
Keywords: insulin resistance; blood glucose; insulin; glucagon; C-peptide; GLP-1; GIP; ghrelin; leptin; PAI-1; resistin; vistatin; adipsin; adiponectin; vagus nerve stimulation; transcutaneous auricular vagus nerve stimulation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Research participants in three groups (normal weight, overweight, obese) will undergo 2 study days (at least one week apart) during which either transcutaneous auricular vagus nerve stimulation (taVNS) or a sham procedure will be performed. The order of the intervention (taVNS or sham procedure) on the two study days is randomized.
Who Masked: Participant
Masking Description: The participants will not be told if transcutaneous auricular vagus nerve stimulation (taVNS) or the sham procedure will be performed. However, it is possible that participants will find out that the stimulation is being performed by a mild tingling sensation associated with taVNS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Normal Weight (Experimental): This arm consists of study participants with a body mass index (BMI) of less than 25. These study participants will participate on two study days. On one study day non-invasive transcutaneous auricular vagus nerve stimulation (taVNS) and on the other study day a sham procedure will be performed. Capillary blood samples (finger prick) will be obtained before and after the interventions on both study days. The ECG will be recorded before, during, and after the intervention on both study days.
  Interventions: Device: taVNS; Device: Sham taVNS
- Overweight (Experimental): This arm consists of study participants with a body mass index (BMI) of more than 25 but less than 30. These study participants will participate on two study days. On one study day non-invasive transcutaneous auricular vagus nerve stimulation (taVNS) and on the other study day a sham procedure will be performed. Capillary blood samples (finger prick) will be obtained before and after the interventions on both study days. The ECG will be recorded before, during, and after the intervention on both study days.
  Interventions: Device: taVNS; Device: Sham taVNS
- Obese (Experimental): This arm consists of study participants with a body mass index (BMI) of more than 30. These study participants will participate on two study days. On one study day non-invasive transcutaneous auricular vagus nerve stimulation (taVNS) and on the other study day a sham procedure will be performed. Capillary blood samples (finger prick) will be obtained before and after the interventions on both study days. The ECG will be recorded before, during, and after the intervention on both study days.
  Interventions: Device: taVNS; Device: Sham taVNS

INTERVENTIONS:
Device: taVNS — A bipolar clip electrode is attached to the auricle at the location of the cymba conchae. Electrical stimulation (30 Hz stimulation frequency, 300 μs pulse width) is applied for 30 min. The stimulation current is determined individually for each participant by slowly increasing the stimulation current until the participants feel a mild tingling sensation at the site of the electrode. Then the current is gradually reduced until the tingling sensation disappears. This current will then be used for taVNS. A TENS 7000 or EMS 7500 device (510(k): K080661) is used.
  Other Names: Transcutaneous Auricular Vagus Nerve Stimulation
Device: Sham taVNS — A bipolar clip electrode is attached to the auricle at the location of the cymba conchae but no electrical current is applied to the electrode.
  Other Names: Sham Transcutaneous Auricular Vagus Nerve Stimulation

SUMMARY:
Being overweight or obese has been associated with insulin resistance contributing to an increased risk for the development of type II diabetes. Food intake, metabolic rate, and blood glucose levels are regulated by the autonomic nervous system, including the vagus nerve. This study evaluates the hypothesis that non-invasive transcutaneous auricular vagus nerve stimulation (taVNS) affects hormones that regulate food intake and blood glucose levels in a way that is consistent with reduced food intake and lower blood glucose levels. The investigators further hypothesize that these effects of taVNS depend on body weight. In a cross-over design generally healthy study participants will receive either taVNS or a sham intervention for 30 minutes on two separate study days. The order of the intervention on the two study days will be randomized and the two study days are at least one week apart. Based on body mass index (BMI) study participants are assigned to either a normal weight (BMI<25), overweight (BMI<30), or obese (BMI>30) group. Capillary blood samples taken by finger prick before and after the intervention on each study day will be analyzed for blood glucose concentration and hormones that are linked to food intake and blood glucose levels. In addition, autonomic function will be assessed by heart rate variability analysis of ECG recordings obtained before, during, and after the intervention on each study day.

DETAILED DESCRIPTION:
Clinical studies and experimental studies in animals have demonstrated that cervical vagus nerve stimulation causes weight loss in obese patients and has profound effects on glucose homeostasis. Furthermore, anorexic and antidiabetic effects have been reported in response to non-invasive transcutaneous auricular vagus nerve stimulation (taVNS). Thus, non-invasive taVNS may potentially prevent insulin resistance in obesity. The objective of this study is to investigate the acute effects of taVNS on hormones and adipokines linking obesity with insulin resistance in human subjects. The hypothesis of this study is that acute application of taVNS elicits anti-diabetic effects through modulation of plasma levels of insulin, glucagon, C-peptide, GLP-1 (stimulates insulin and suppresses glucagon release), and GIP (gastric inhibitory polypeptide, stimulates insulin secretion). Furthermore, the investigators hypothesize that taVNS elicits anorexic effects by modulating ghrelin and leptin plasma levels. Finally the investigators hypothesize that taVNS may reduce the impact of obesity on insulin resistance by modulating PAI-1 (plasminogen activator inhibitor-1; increased in obesity and metabolic syndrome), resistin (adipose tissue secretory factor, suggested to link obesity with insulin resistance), vistatin (enriched in visceral fat and may stimulate the insulin receptor), adipsin (secreted from adipocytes; improves β-cell function), and adiponectin (secreted from adipose tissue; increases insulin sensitivity). In normal weight (BMI<25, n=14), overweight (BMI<30, n=14), and obese (BMI>30, n=14) and otherwise healthy study participants blood glucose levels and plasma concentrations (finger prick blood sampling) of insulin, glucagon, C-peptide, GLP-1, GIP, ghrelin, leptin, PAI-1, resistin, vistatin (Bio-Plex kit 171A7001M), adipsin, and adiponectin (Bio-Plex kit 171A7002M) will be determined before and after 30 minutes of taVNS (EMS 7500, 10 Hz, 300ms, n=7 in each body weight group) or sham taVNS (control experiment, n=7 in each body weight group). Before, during and after taVNS or sham taVNS autonomic function will be assessed by heart rate variability analysis from ECG recordings. The investigators expect that the outcome of this study will demonstrate that taVNS lowers blood glucose levels and elicits hormone/adipokine responses consistent with anorexia and improved insulin resistance. The investigators further hypothesize that these effects of taVNS will be more pronounced in obese compared to overweight and normal weight study participants.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy

Exclusion Criteria:

* Age under 18 years
* Pregnancy
* Acute illnesses/fever
* Any medication that interferes with the autonomic nervous system (e.g., beta blockers)
* Any medication that interferes with glucose metabolism (e.g., antidiabetic drugs)
* Any medication that interferes with lipid metabolism (e.g., statins)
* Any medical conditions that interfere with the autonomic nervous system
* Type 1 or Type 2 diabetes
* Epilepsy
* Cardiac conditions, including arrhythmia
* Vestibulocochlear neuronitis or nerve damage (e.g., hearing loss or tinnitus)
* Skin irritation/inflammation at the stimulation site at the ear
* Current drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-04-26 (Actual)

PRIMARY OUTCOMES:
Change in Blood Glucose Concentration induced by taVNS | During the taVNS intervention (30 min).
  The blood glucose concentration is measured before and after application of taVNS from capillary blood samples obtained by finger prick. The change in blood glucose concentration is determined as the difference in the two blood glucose concentrations (after taVNS minus before taVNS).
Change in Blood Glucose Concentration induced by sham taVNS | During the sham taVNS intervention (30 min).
  The blood glucose concentration is measured before and after application of sham taVNS from capillary blood samples obtained by finger prick. The change in blood glucose concentration is determined as the difference in the two blood glucose concentrations (after sham taVNS minus before sham taVNS).
Change in Insulin Plasma Concentration induced by taVNS | During the taVNS intervention (30 min).
  Using capillary blood samples obtained by finger prick the insulin plasma concentration will be determined using a Bioplex assay. The insulin plasma concentration will be determined before and after application of taVNS and the change in plasma concentration will be determined as the difference in the plasma concentrations (after taVNS minus before taVNS).
Change in Insulin Plasma Concentration induced by sham taVNS | During the taVNS intervention (30 min).
  Using capillary blood samples obtained by finger prick the insulin plasma concentration will be determined using a Bioplex assay. The insulin plasma concentration will be determined before and after application of sham taVNS and the change in plasma concentration will be determined as the difference in the plasma concentrations (after sham taVNS minus before sham taVNS).
Change in Glucagon Plasma Concentration induced by taVNS | During the taVNS intervention (30 min).
  Using capillary blood samples obtained by finger prick the glucagon plasma concentration will be determined using a Bioplex assay. The glucagon plasma concentration will be determined before and after application of taVNS and the change in plasma concentration will be determined as the difference in the plasma concentrations (after taVNS minus before taVNS).
Change in Glucagon Plasma Concentration induced by sham taVNS | During the taVNS intervention (30 min).
  Using capillary blood samples obtained by finger prick the glucagon plasma concentration will be determined using a Bioplex assay. The glucagon plasma concentration will be determined before and after application of sham taVNS and the change in plasma concentration will be determined as the difference in the plasma concentrations (after sham taVNS minus before sham taVNS).
Change in C-Peptide Plasma Concentration induced by taVNS | During the taVNS intervention (30 min).
  Using capillary blood samples obtained by finger prick the C-peptide plasma concentration will be determined using a Bioplex assay. The C-peptide plasma concentration will be determined before and after application of taVNS and the change in plasma concentration will be determined as the difference in the plasma concentrations (after taVNS minus before taVNS).
Change in C-Peptide Plasma Concentration induced by sham taVNS | During the taVNS intervention (30 min).
  Using capillary blood samples obtained by finger prick the C-peptide plasma concentration will be determined using a Bioplex assay. The C-peptide plasma concentration will be determined before and after application of sham taVNS and the change in plasma concentration will be determined as the difference in the plasma concentrations (after sham taVNS minus before sham taVNS).
Change in GLP-1 Plasma Concentration induced by taVNS | During the taVNS intervention (30 min).
  Using capillary blood samples obtained by finger prick the GLP-1 plasma concentration will be determined using a Bioplex assay. The GLP-1 plasma concentration will be determined before and after application of taVNS and the change in plasma concentration will be determined as the difference in the plasma concentrations (after taVNS minus before taVNS).
Change in GLP-1 Plasma Concentration induced by sham taVNS | During the taVNS intervention (30 min).
  Using capillary blood samples obtained by finger prick the GLP-1 plasma concentration will be determined using a Bioplex assay. The GLP-1 plasma concentration will be determined before and after application of sham taVNS and the change in plasma concentration will be determined as the difference in the plasma concentrations (after sham taVNS minus before sham taVNS).
Change in GIP Plasma Concentration induced by taVNS | During the taVNS intervention (30 min).
  Using capillary blood samples obtained by finger prick the GIP plasma concentration will be determined using a Bioplex assay. The GIP plasma concentration will be determined before and after application of taVNS and the change in plasma concentration will be determined as the difference in the plasma concentrations (after taVNS minus before taVNS).
Change in GIP Plasma Concentration induced by sham taVNS | During the taVNS intervention (30 min).
  Using capillary blood samples obtained by finger prick the GIP plasma concentration will be determined using a Bioplex assay. The GIP plasma concentration will be determined before and after application of sham taVNS and the change in plasma concentration will be determined as the difference in the plasma concentrations (after sham taVNS minus before sham taVNS).
Change in Ghrelin Plasma Concentration induced by taVNS | During the taVNS intervention (30 min).
  Using capillary blood samples obtained by finger prick the ghrelin plasma concentration will be determined using a Bioplex assay. The ghrelin plasma concentration will be determined before and after application of taVNS and the change in plasma concentration will be determined as the difference in the plasma concentrations (after taVNS minus before taVNS).
Change in Ghrelin Plasma Concentration induced by sham taVNS | During the taVNS intervention (30 min).
  Using capillary blood samples obtained by finger prick the ghrelin plasma concentration will be determined using a Bioplex assay. The ghrelin plasma concentration will be determined before and after application of sham taVNS and the change in plasma concentration will be determined as the difference in the plasma concentrations (after sham taVNS minus before sham taVNS).
Change in Leptin Plasma Concentration induced by taVNS | During the taVNS intervention (30 min).
  Using capillary blood samples obtained by finger prick the leptin plasma concentration will be determined using a Bioplex assay. The leptin plasma concentration will be determined before and after application of taVNS and the change in plasma concentration will be determined as the difference in the plasma concentrations (after taVNS minus before taVNS).
Change in Leptin Plasma Concentration induced by sham taVNS | During the taVNS intervention (30 min).
  Using capillary blood samples obtained by finger prick the leptin plasma concentration will be determined using a Bioplex assay. The leptin plasma concentration will be determined before and after application of sham taVNS and the change in plasma concentration will be determined as the difference in the plasma concentrations (after sham taVNS minus before sham taVNS).
Change in PAI-1 Plasma Concentration induced by taVNS | During the taVNS intervention (30 min).
  Using capillary blood samples obtained by finger prick the PAI-1 plasma concentration will be determined using a Bioplex assay. The PAI-1 plasma concentration will be determined before and after application of taVNS and the change in plasma concentration will be determined as the difference in the plasma concentrations (after taVNS minus before taVNS).
Change in PAI-1 Plasma Concentration induced by sham taVNS | During the taVNS intervention (30 min).
  Using capillary blood samples obtained by finger prick the PAI-1 plasma concentration will be determined using a Bioplex assay. The PAI-1 plasma concentration will be determined before and after application of sham taVNS and the change in plasma concentration will be determined as the difference in the plasma concentrations (after sham taVNS minus before sham taVNS).
Change in Resistin Plasma Concentration induced by taVNS | During the taVNS intervention (30 min).
  Using capillary blood samples obtained by finger prick the resistin plasma concentration will be determined using a Bioplex assay. The resistin plasma concentration will be determined before and after application of taVNS and the change in plasma concentration will be determined as the difference in the plasma concentrations (after taVNS minus before taVNS).
Change in Resistin Plasma Concentration induced by sham taVNS | During the taVNS intervention (30 min).
  Using capillary blood samples obtained by finger prick the resistin plasma concentration will be determined using a Bioplex assay. The resistin plasma concentration will be determined before and after application of sham taVNS and the change in plasma concentration will be determined as the difference in the plasma concentrations (after sham taVNS minus before sham taVNS).
Change in Vistatin Plasma Concentration induced by taVNS | During the taVNS intervention (30 min).
  Using capillary blood samples obtained by finger prick the vistatin plasma concentration will be determined using a Bioplex assay. The vistatin plasma concentration will be determined before and after application of taVNS and the change in plasma concentration will be determined as the difference in the plasma concentrations (after taVNS minus before taVNS).
Change in Vistatin Plasma Concentration induced by sham taVNS | During the taVNS intervention (30 min).
  Using capillary blood samples obtained by finger prick the vistatin plasma concentration will be determined using a Bioplex assay. The vistatin plasma concentration will be determined before and after application of sham taVNS and the change in plasma concentration will be determined as the difference in the plasma concentrations (after sham taVNS minus before sham taVNS).
Change in Adipsin Plasma Concentration induced by taVNS | During the taVNS intervention (30 min).
  Using capillary blood samples obtained by finger prick the adipsin plasma concentration will be determined using a Bioplex assay. The adipsin plasma concentration will be determined before and after application of taVNS and the change in plasma concentration will be determined as the difference in the plasma concentrations (after taVNS minus before taVNS).
Change in Adipsin Plasma Concentration induced by sham taVNS | During the taVNS intervention (30 min).
  Using capillary blood samples obtained by finger prick the adipsin plasma concentration will be determined using a Bioplex assay. The adipsin plasma concentration will be determined before and after application of sham taVNS and the change in plasma concentration will be determined as the difference in the plasma concentrations (after sham taVNS minus before sham taVNS).
Change in Adiponectin Plasma Concentration induced by taVNS | During the taVNS intervention (30 min).
  Using capillary blood samples obtained by finger prick the adipsin plasma concentration will be determined using a Bioplex assay. The adiponectin plasma concentration will be determined before and after application of taVNS and the change in plasma concentration will be determined as the difference in the plasma concentrations (after taVNS minus before taVNS).
Change in Adiponectin Plasma Concentration induced by sham taVNS | During the taVNS intervention (30 min).
  Using capillary blood samples obtained by finger prick the adipsin plasma concentration will be determined using a Bioplex assay. The adiponectin plasma concentration will be determined before and after application of sham taVNS and the change in plasma concentration will be determined as the difference in the plasma concentrations (after sham taVNS minus before sham taVNS).

SECONDARY OUTCOMES:
Changes in Autonomic Function induced by taVNS | During the taVNS intervention (30 min).
  Autonomic function will be assessed by heart rate variability analysis of ECG recordings obtained before and after application of taVNS. Changes in autonomic function will be determined by the difference in heart rate variability before and after taVNS (after taVNS minus before taVNS).
Changes in Autonomic Function induced by sham taVNS | During the sham taVNS intervention (30 min).
  Autonomic function will be assessed by heart rate variability analysis of ECG recordings obtained before and after application of sham taVNS. Changes in autonomic function will be determined by the difference in heart rate variability before and after sham taVNS (after sham taVNS minus before sham taVNS).

CONTACTS AND LOCATIONS:
Overall Officials: Harald M Stauss, MD, PhD, Principal Investigator — Burrell College of Osteopathic Medicine
Locations (1):
- Burrell College of Osteopathic Medicine, Las Cruces, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No